CLINICAL TRIAL: NCT01805115
Title: A Randomized Comparison of Oral, Sublingual and Vaginal Misoprostol Administration in Premenopausal Women Before Operative Hysteroscopy
Brief Title: Misoprostol Administration Before Operative Hysteroscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, CHA University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KNC13-005
Record Dates: First submitted 2013-03-04; First posted 2013-03-06 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Endometrial Disorder
Keywords: hysteroscopy; misoprostol
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oral misoprostol (Experimental): The oral group (misoprostol 400 ug) self-administered the medications orally 8-10 h before surgery.
  Interventions: Drug: Oral misoprostol
- Sublingual misoprostol (Experimental): The sublingual group (misoprostol 400 ug) self-administered the medications sublingually 8-10 h before surgery.
  Interventions: Drug: Sublingual misoprostol
- Vaginal misoprostol (Experimental): The vaginal group (misoprostol 400 ug) self-administered the medications vaginally 8-10 h before surgery.
  Interventions: Drug: Vaginal misoprostol
- Control (Experimental): The no-misoprostol group did not administer the medication of misoprostol before the procedure
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Oral misoprostol — Patients were randomly allocated at the outpatient department into 4 groups with a ratio of 1:1:1:1: the oral, sublingual, vaginal, and no misoprostol group received all 400 μg of misoprostol (two tablets of Cytotec; 200 μg). All misoprostol tablets were identical and patients were blinded to group allocation
  Other Names: two tablets of Cytotec (200 μg)
  Arms: Oral misoprostol
Drug: Sublingual misoprostol — Patients were randomly allocated at the outpatient department into 4 groups with a ratio of 1:1:1:1: the oral, sublingual, vaginal, and no misoprostol group received all 400 μg of misoprostol (two tablets of Cytotec; 200 μg). All misoprostol tablets were identical and patients were blinded to group allocation
  Other Names: two tablets of Cytotec (200 μg)
  Arms: Sublingual misoprostol
Drug: Vaginal misoprostol — Patients were randomly allocated at the outpatient department into 4 groups with a ratio of 1:1:1:1: the oral, sublingual, vaginal, and no misoprostol group received all 400 μg of misoprostol (two tablets of Cytotec; 200 μg). All misoprostol tablets were identical and patients were blinded to group allocation
  Other Names: two tablets of Cytotec (200 μg)
  Arms: Vaginal misoprostol
Drug: Control — The control group was not given any cervical priming agents or placebo.
  Arms: Control

SUMMARY:
The objective of this study is to compare the efficacy of oral, sublingual, vaginal, and no misoprostol prior to operative hysteroscopy in premenopausal women.

DETAILED DESCRIPTION:
The route of administration of misoprostol for cervical dilatation prior to operative hysteroscopy can be oral, vaginal, or sublingual. However, it is still unclear which route is more effective and less harmful for cervical dilation prior to operative hysteroscopy in premenopausal women. Furthermore, there have been no studies comparing among oral, sublingual, and vaginal misoprostol, no medication (control) in these women. The objective of this study is to compare the efficacy and safety of oral, sublingual, vaginal, and no misoprostol prior to operative hysteroscopy in premenopausal women.

ELIGIBILITY:
Inclusion Criteria:

Symptomatic patients that were suspected as having intrauterine pathology, such as submucosal myoma, endometrial polyp or other endometrial pathological findings based on the transvaginal ultrasound, were enrolled.

Inclusion criteria were as follows: women who were of reproductive age (i.e., were premenopausal) and were not pregnant at the time of presentation (i.e., negative for urine pregnancy test or last menstrual period within the last 4 weeks). -

Exclusion Criteria:

Exclusion criteria included any evidence of a contraindication to prostaglandins (history of severe asthma, glaucoma, preexisting severe cardiac disease, or renal failure), or allergy to prostaglandins, any sign of genital infection, presence of significant uterovaginal prolapse that could affect administration of vaginal tablets, history of cervical surgery, presence of space occupying lesions in endocervical canal, and treatment of GnRH agonist.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
the preoperative cervical width | just before the operation (From finish of anesthesic induction to introduction of a rigid resectoscope with 10-mm outer sheath diameter in uterine cavity)
  The primary outcome measure was the preoperative cervical width at the time of operation. The cervical width was assessed by performing cervical dilation, starting with a number 10 Hegar dilator and subsequently inserting smaller Hegar dilators until dilator could pass through the internal os without resistance. The largest one that could be passed was recorded as the initial cervical width.

SECONDARY OUTCOMES:
misoprostol-associated side effects | before the procedures

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD, Principal Investigator — Department of Obstetrics and Gynecology, CHA Gangnam Medical Center, CHA University, Seoul, Korea
Locations (1):
- CHA Gangnam Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Song T, Kim MK, Kim ML, Jung YW, Yoon BS, Seong SJ. Effectiveness of different routes of misoprostol administration before operative hysteroscopy: a randomized, controlled trial. Fertil Steril. 2014 Aug;102(2):519-24. doi: 10.1016/j.fertnstert.2014.04.040. Epub 2014 May 23. PMID 24856464